CLINICAL TRIAL: NCT02644889
Title: Epidermal Growth Factor Receptor (EGFR) Mutation Detection From Advanced Non-small Cell Lung Cancer Tissue and Plasma in Tyrosine Kinase Inhibitor (TKI) Treatment
Brief Title: EGFR Mutation Detection From Advanced NSCLC Patient Tissue and Plasma in EGFR-TKI Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GenoSaber (Industry)
Responsible Party: Sponsor
Other Study IDs: EGFR2015-02
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Epidermal growth factor receptor(EGFR); NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients advanced NSCLC EGFR mutated: This is an observational study, there is no intervention.

SUMMARY:
This study has been designed in order to detect EGFR mutation abundance of tissue and concentration of plasma from Advanced Non-small Cell Lung Cancer during treatment with Tyrosine Kinase Inhibitor (TKI) .Through this experiment the investigators aim to evaluate the feasibility of plasma EGFR detection and evaluate the correlation of EGFR mutations and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years and under 75 years
* Histologically and cytologically proven non-small Cell Lung Cancer
* Clinical stages Ⅲ ~ Ⅳ
* Not receive any anti-tumor treatment
* Eastern cooperative oncology group performance status (ECOG PS) =1~2
* Estimated survival time more than 3 months
* EGFR-TKI treatment for first-line or second-line
* Voluntary to participate in this clinical trial and sign the consent form

Exclusion Criteria:

* Patients have received EGFR-TKI therapy before the study
* With other malignancy history in the recent 5 years before the study
* Pregnancy or breast feeding phase
* Inadequate samples for testing
* Follow-up compliance is poor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage Ⅲ-Ⅳ NSCLC with EGFR mutations and who began a treatment by TKI .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
EGFR Mutation Detection of FFPE and plasma samples | baseline
  To evaluate the feasibility of plasma EGFR detection from non-small cell lung cancer patients harboring EGFR activating mutation who are being treated with EGFR TKIs and evaluate the correlation of EGFR mutations and prognosis.
EGFR Mutation Detection of plasma samples for the following-up patients who take TKI. | From start of treatment to time of progression or death, whichever occurs first, assessed up to 3 years
  In order to monitor the change of plasma EGFR mutation copy number.